CLINICAL TRIAL: NCT01700855
Title: Electroacupuncture for Pain Relief in Patients With Nasal Sinus Surgery and Mammaplasty: a Randomized Controlled Study
Brief Title: Electroacupuncture Anesthesia for Nasal Sinus Surgery and Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, wangqiang, Associate Professor, Associate Consultant, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mazuike-28
Record Dates: First submitted 2012-09-03; First posted 2012-10-04 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2012-05

CONDITIONS: Therapeutic (Nonsurgical) and Rehabilitative Anesthesiology Devices Associated With Adverse Incidents
Keywords: Electroacupuncture; Analgesia; Anesthesia; Nasal septoplasty; Mammaplasty
MeSH Terms: conditions — Agnosia | interventions — salicylhydroxamic acid; Electroacupuncture; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture (Experimental): Patients received electroacupuncture stimulation
  Interventions: Procedure: Electroacupuncture
- Non-electroacupuncture (Sham Comparator): Patients received sham electroacupuncture
  Interventions: Procedure: non-electroacupuncture

INTERVENTIONS:
Procedure: non-electroacupuncture — The same procedure as electroacupuncture except stimulation
  Other Names: Sham
  Arms: Non-electroacupuncture
Procedure: Electroacupuncture — Electrodes are applied to bilateral "Hegu(L14)" acupoints at the time of 1h before operation, and connected to Hwato Electronic Acupuncture Treatment Instrument (Model No. SDZ-V, Suzhou Medical Appliances Co., Ltd., Suzhou, China). The acupoints are stimulated at an intensity of 3~6 mA and a frequency of 2/30 Hz for 30 min. The highest intensity will be chosen at which the patient can tolerate.
  Other Names: Electroacupuncture preconditioning; Electroacupuncture pretreatment; Transcutaneous electric nerve stimulation
  Arms: Electroacupuncture

SUMMARY:
The purpose of this study is to verify the intraoperative analgesia of electroacupuncture in patients undergoing selective nasal sinus surgery and mammaplasty.

DETAILED DESCRIPTION:
Acupuncture therapy has been proved helpful in the patients suffering from various pain problems. And it is reported to be able to reduce the intraoperative anesthetic requirement. However, so far there is few evidence from randomized controlled studies to confirm the assistant anesthetic effect of acupuncture. Electroacupuncture (EA) is a modern non-invasive technique of traditional acupuncture. Compared to traditional acupuncture, EA is more practicable, more easily to be accepted by patients and operated by physicians. Nasal sinus surgery and mammaplasty, especially breast augmentation, mostly belong to the scope of day surgeries, which demand a rapid, smooth recovery from anesthesia with minimum adverse side effects (e.g.: pain, PONV, etc).

ELIGIBILITY:
Inclusion Criteria:

* selective nasal sinus surgery
* selective mammaplasty
* patients who accept the follow-up and sign the informed consent
* ASA 1~2

Exclusion Criteria:

* emergent surgery
* pregnant or breast-feeding women
* coagulopathy
* history of gastrointestinal ulcer
* liver or renal dysfunction
* enrollment in other clinical trials at the same time not reaching the primary endpoint and probably interference the present trial

Ages: 29 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the mean infusion rate of intraoperative remifentanil and propofol | during operation
  To investigate the operative time and total volume of remifentanil and propofol used during operation, and then calculate the mean infusion rate. To assess whether intraoperative requirements for anesthetic drugs could be reduced by EA pretreatment.

SECONDARY OUTCOMES:
Visual analogue scale | post-operative 4h, 8h, 24h and 48h
  To assess whether EA pretreatment could help in alleviating acute post-operative pain.
Extubation time | postoperation
  To investigate the time from the end of propofol and remifentanil infusion to extubation. To assess whether EA pretreatment could shorten the extubation time.

OTHER OUTCOMES:
plasma β-endorphin and cortisol concentration | preoperation, 0h and 24h postoperation
  To assess whether EA pretreatment could increase the plasma levels of β-endorphin and cortisol.
Ramsay score | post-operative 4h, 8h, 24h, 48h
  To assess the effect of EA pretreatment on post-operative Ramsay scores.
incidence of post-operative nausea and vomiting (PONV) | within post-operative 24 hours
  To assess the effect of EA pretreatment on PONV.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, M.D., Ph.D., Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Wang H, Xie Y, Zhang Q, Xu N, Zhong H, Dong H, Liu L, Jiang T, Wang Q, Xiong L. Transcutaneous electric acupoint stimulation reduces intra-operative remifentanil consumption and alleviates postoperative side-effects in patients undergoing sinusotomy: a prospective, randomized, placebo-controlled trial. Br J Anaesth. 2014 Jun;112(6):1075-82. doi: 10.1093/bja/aeu001. Epub 2014 Feb 26. PMID 24576720